CLINICAL TRIAL: NCT06617754
Title: InternatioNal seVerE CRSwNP Registry (INVENT) 2024-2028
Brief Title: International Severe CRSwNP Registry 2024-2028
Acronym: INVENT
Status: Active, not recruiting | Type: Observational
Sponsor: Vibeke Backer (Other)
Collaborators: The European Forum for Research and Education in Allergy and Airway Diseases (Other)
Responsible Party: Sponsor-Investigator, Vibeke Backer, MD, DMSci, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-21020685
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Keywords: CRSwNP; Asthma; Biologic treatment; Effect of treatment; Different geographic collection
MeSH Terms: conditions — Asthma | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (13):
- Patients from Danish registry of global airways: Patients included in the Danish Global Airways Registry
  Interventions: Biological: Biologic drugs
- Patients from the Belgian registry of global airways: Patients included in the Belgian Global Airways Registry
  Interventions: Biological: Biologic drugs
- Patients from the Netherlands registry of global airways: Patients included in the Netherlands registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from the German registry of global airways: Patients included in the German registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from the Swiss registry of global airways: Patients included in the Swiss registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from the Italian registry of global airways: Patients included in the Italian registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from the Portuguese registry of global airways: Patients included in the Portuguese registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from the Finnish registry of global airways: Patients included in the Finnish registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from the US registry of global airways: Patients included in the US registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from the Australian registry of global airways: Patients included in the Australian registry of global airways
  Interventions: Biological: Biologic drugs
- Patients from Spanish registry of global airways: Patients included in the Spanish Global Airways Registry
- Patients from Polish registry of global airways: Patients included in the Polish Global Airways Registry
  Interventions: Biological: Biologic drugs
- Patients from French registry of global airways: Patients included in the French Global Airways Registry
  Interventions: Biological: Biologic drugs

INTERVENTIONS:
Biological: Biologic drugs — Biologic drugs including Mepolizumab, Dupilumab, Omalizumab, Tezepelumab, or future monoclonal antibodies
  Groups: Patients from Danish registry of global airways; Patients from French registry of global airways; Patients from Polish registry of global airways; Patients from the Australian registry of global airways; Patients from the Belgian registry of global airways; Patients from the Finnish registry of global airways; Patients from the German registry of global airways; Patients from the Italian registry of global airways; Patients from the Netherlands registry of global airways; Patients from the Portuguese registry of global airways; Patients from the Swiss registry of global airways; Patients from the US registry of global airways

SUMMARY:
The objective of the study is to collect real-life data worldwide, which already have been collected in national databases, to merge the data and the knowledge with the focus of better care for the individual patients, more efficient use of the hospital cost of biologics and working for "personalized medicine".

DETAILED DESCRIPTION:
Regional or national registries have evaluated the efficacy of different biologics in severe uncontrolled CRSwNP coordinated by several academic centres in Europe. At present, these registries have not been merged nor allowed the comparison in real-life efficacy between the 3 different monoclonal antibodies (mepolizumab, dupilumab, omalizumab) with different mechanism which has been approved for the indication of CRSwNP and the effect of the nasal polyp score. Some countries have allowance for some of the different biologic drugs, other countries have other combination of the drugs. Despite the heterogeneity in availability of biologics for the indication of CRSwNP, the merge of data might lead to very interesting outcomes.

The objective of the study is to collect real-life data worldwide, which already have been collected in national databases, to merge the data and the knowledge with the focus of better care for the individual patients, more efficient use of the hospital cost of biologics and working for "personalized medicine".

Compare the outcomes of different biologics in different national registries, at screening and 6-month follow-up: Primary aims:

1. Delphi process to point at the viable of importance.
2. The speed and size of SNOT-22 reduction
3. The speed and size of NPS reduction
4. The speed and size of Nasal congestion score (NCS) reduction
5. The speed and size of smell score increase.
6. The CTscan/Lund-Mackay score response
7. The evolution of the response on VAS scale (patients)
8. The Type 2 biomarkers at entrance and during the study
9. The (non)responder percentages defined based on EUFOREA criteria
10. The use of OCS (amount and frequency)
11. The frequency and time (days) since last sinus surgery
12. The effect of biologics on comorbidities (atopic dermatitis, allergic rhinitis, asthma and NSAID intolerance) in patients with CRSwNP
13. The reduced in need of Otrivin or similar drugs
14. Differences between inclusion criteria for biologic drugs, and differences between countries.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of CRSwNP
* Indication for biologic treatment as suggested by EPOS/EUFOREA
* Have been followed for 6 months

Exclusion Criteria:

* Unilateral polyps
* Non-Type-2 inflammation
* Treatment less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In Denmark, the study population consists of patients suffering CRSwNP and treated with biologic treatments included in global airways Danish/National registry.
  In the other countries, the study population consists of patients suffering CRSwNP and treated with biologic treatments who are included in local Registries.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Change in The Sino-Nasal Outcome Test 22 (SNOTT22) score | 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, and 60 months follow up
  The success rate indicated by a significant change in health-related quality of life related to nasal symptoms measured with the questionnaire SNOT22.
Change in Nasal Polyp Score (NPS) | 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, and 60 months follow up
  The NPS scale ranges from 0 (no polyp) to 4 (large polyps) for each nostril. The total score ranging from 0-8.
Change in visual analogue scale (VAS) | 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, and 60 months follow up
  Change in VAS related to nasal symptoms. Minimum score = 0 and maximum score = 10. High score indicates worse nasal symptoms
Change in olfactory function | 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, and 60 months follow up
  Change in olfactory function measured with Sniffin' Stick 16 blue. Minimum score = 0. Maximum score = 16. A score between 0-8 indicates anosmia, a score between 8-11 indicates hyposmia, and a score >11 indicates normosmia.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rhinolaryngology Head & Neck surgery and Audiology, Copenhagen, Denmark, Denmark